CLINICAL TRIAL: NCT05874583
Title: Prevention of Bleeding in Total Joint Replacement: Contribution of Combined Route in Tranexamic Acid Administration
Brief Title: Prevention of Bleeding in Total Joint Replacement: Combined Route Administration of Tranexamic Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TXA in joint replacement
Record Dates: First submitted 2023-04-26; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Tranexamic Acid; Arthroplasty, Replacement, Knee; Blood Transfusion; Arthroplasty, Replacement, Hip
MeSH Terms: interventions — Administration, Topical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Group (Active Comparator): patients receiving 2 doses of 1 g of tranexamic acid in in intra venous route 3 hours apart
  Interventions: Drug: Intravenous route Tranexamic acid injection
- Combined Group (Experimental): receiving the first 1g of tranexamic acid Intra venously and the second topical dose was 1,5g after reduction of the fascia.
  Interventions: Drug: Combined route administration of Tranexamic acid

INTERVENTIONS:
Drug: Combined route administration of Tranexamic acid — tranexamic acid in topical route administration
  Other Names: Intravenous and topical administration
  Arms: Combined Group
Drug: Intravenous route Tranexamic acid injection — Intra venous route administration
  Other Names: Intravenously only
  Arms: Intravenous Group

SUMMARY:
The investigators aimed to compare two doses of intravenous (IV) tranexamic acid (TXA) with a combined single dose of topical and IV TXA on haemoglobin decline 24 hours after total joint arthroplasties.

The investigators conducted randomized, double-blind trial. The participants were randomized to either intrvenous group receiving 2 doses of 1 gram TXA in intravenous route 3 hours apart, or a combined application group receiving the first 1 gram IV and the topical dose was 1.5 gram after reduction of the fascia.

DETAILED DESCRIPTION:
The investigators provided the pre-anaesthetic consultation. They carried out a rigorous clinical examination, a balancing of the defects and an adjustment of the therapies. The patients' written and informed consent was obtained. All patients had a preoperative blood count, blood grouping, renal assessment with dosage of uremia and creatinine. The investigators calculated the tolerable losses (mL). Randomization and allocation were carried out at this stage by an anesthesiologist other than the one managing the patient perioperatively.

On arrival in the operating room, the investigators set up the following systematic monitoring: electrocardioscope, pulse oximetry, gas analyzer, monitoring of capnia and curarization in the event of general anesthesia, non-invasive blood pressure. Two peripheral venous approaches were put in place. All patients received antibiotic prophylaxis with 2 g of Cefazolin and in case of allergy 900 mg of Dalacin. The anesthetic protocol was standardized. The choice between general or locoregional anesthesia was left to the discretion of the anesthesiologist treating the patient. For each patient, the investigators specified: The surgical approach, the type of prosthesis (cemented or not), the intraoperative posture, the duration of the procedure and of the anesthesia. During intraoperative monitoring, any hypotension with a decrease in mean arterial pressure of 20% of the baseline value for a period of more than 3 minutes or other complications were mentioned. The estimated bleeding (contents of the suction jar, number of drapes and compresses soaked in blood) with determination of the percentage of total losses intraoperatively as well as the results of the intraoperative blood count (if deemed necessary) were also specified. Transfusion of labile blood products was managed according to the patient's terrain, the degree of anemia, the speed of onset of the anemia and his hemodynamic tolerance. The analgesic protocol was also standardized.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged of 18 years or more;
* Primary total hip or knee arthroplasty;
* A traumatic, degenerative or malformative setting.

Exclusion Criteria:

* Revisions;
* Bilateral procedures;
* Polytrauma;
* Pregnant patients;
* Contraindications for the use of TXA, Coagulation disorders or anaemia with Haemoglobin (Hb) less than or equal to 9 g/dl preoperatively;
* Patients treated with anticoagulants, Heparin, Warfarin, Oestrogen.
* Serious anaesthesia-related complications (impossible orotracheal intubation , anaphylactic shock);
* Severe transfusion reaction such as haemolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Haemoglobin decline | up to 24 hours after surgery
  The decline of hemoglobin levels

SECONDARY OUTCOMES:
The use of blood transfusion | up to 24 hours after surgery.
  Number of transfusion needed

OTHER OUTCOMES:
Thromboembolic complications | Up to 3 months after surgery
  postoperative deep vein thrombosis or pulmonary embolism

CONTACTS AND LOCATIONS:
Overall Officials: Mhamed Sami MS Mebazaa, Pr, Principal Investigator — Mongi Slim local research ethical committee
Locations (1):
- Mongi Slim University Hospital, La Marsa, Tunis Governorate, Tunisia